CLINICAL TRIAL: NCT05030259
Title: ACS After Femoropopliteal Arterial Injuries
Brief Title: The Research About the ACS After Femoropopliteal Arterial Injuries
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HZY005ACS
Record Dates: First submitted 2021-08-03; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Acute Compartment Syndrome
Keywords: ACS; femoropopliteal arterial injuries; fasciotomy
MeSH Terms: interventions — Fasciotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with fasciotomy
  Interventions: Procedure: fasciotomy
- patients without fasciotomy

INTERVENTIONS:
Procedure: fasciotomy — To perform fasciotomy
  Groups: patients with fasciotomy

SUMMARY:
Crural Compartment syndrome is a well-known sequela after femoropopliteal arterial injuries in the lower extremity, particularly when there has been a long period of ischemia,need for ligation of a major vein, or when there is severe associated soft tissue.There is conteoversy in the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with femoropopliteal arterial injuries
* patients older than 18 years

Exclusion Criteria:

* Patients who did not survive to discharge
* Patients with primary amputation
* patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with femoropopliteal arterial injuries in our hospital who will be treated with vascular repair.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of amputation | up to 6 months
fasciotomy performed or not | up to 2 weeks

SECONDARY OUTCOMES:
the rate of primary skin closure | up to 1 months
hospital lengths of stay | up to 6 months
injury mechanism of patients | up to 1 week
the costs of hospitalization | up to 2 months
tourniquet used or not | up to 1 week
the time of using tourniquet | up to 1 week
the time to surgical intervention | up to 1 month
extremity Abbreviated Injury Scale of patients | up to 1 week
  minimum is 1, maximum is 6, higher scores mean a worse outcome
Injury Severity Score of patients | up to 1 week
  minimum is 0, maximum is 75, higher scores mean a worse outcome
concomitant injury of patients | up to 1 week
time of skin closure | up to 1 month
admission hemoglobin of patients | up to 1 month
admission pH of patients | up to 1 month
admission lactate of patients | up to 1 month
postoperative lactate of patients | up to 1 month
admission International Normalized Ratio of patients | up to 1 month
postoperative International Normalized Ratio of patients | up to 1 month
admission CK of patients | up to 1 month
postoperative CK of patients | up to 1 month
admission LDH of patients | up to 1 month
postoperative LDH of patients | up to 1 month
Number of Participants with Lower Extremity Arteriosclerosis Obliterans | up to 1 week
vascular repair technique of patients | up to 1 week
Number of Participants with sepsis | up to 1 month
Ischemia time of patients | up to 1 week
Postoperative knee function of patients | up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hou Zhiyong, Doctor, Principal Investigator — Hebei Medical University Third Hospital
Locations (1):
- the Third Hospital of Hebei Medical Univesity, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
acute compartment syndrome
Supporting Information: Study Protocol
Time Frame: 2 years after the experiment was conducted
Access Criteria: all authors focusing on ACS research